CLINICAL TRIAL: NCT00329303
Title: Follow-up of Study C87040: Multicentre, Double-blind Study to Describe the Efficacy and Safety of Re-treatment With CDP870 (Certolizumab Pegol) Subcutaneous at 2 Different Dose Regimens (400 mg Initial Dose at Week 0 With 200 mg Every 2 Weeks Thereafter and 400 mg Every 2 Weeks) or Placebo for 12 Weeks, in Subjects Suffering From Moderate-to-severe Chronic Plaque Psoriasis Who Are Candidates for Systemic Therapy and/or Phototherapy and/or Photochemotherapy, Having Responded to Treatment in Study C87040 and Having Subsequently Relapsed
Brief Title: Efficacy of Re-treatment With Cimzia® in Subject With Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C87044; 2005-005525-63 (EudraCT Number)
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-02

CONDITIONS: Psoriasis
Keywords: Moderate to severe chronic plaque psoriasis; anti TNF α; CDP 870; Cimzia®; certolizumab pegol; retreatment
MeSH Terms: conditions — Psoriasis | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Certolizumab Pegol (CZP) 200 mg (Experimental): Subcutaneous injections of 400 mg initial dose at Week 0 with 200 mg every 2 weeks thereafter.
  Interventions: Drug: Certolizumab Pegol (Cimzia®)
- Certolizumab Pegol (CZP) 400 mg (Experimental): Subcutaneous injections of 400 mg every 2 weeks.
  Interventions: Drug: Certolizumab Pegol (Cimzia®)

INTERVENTIONS:
Drug: Certolizumab Pegol (Cimzia®) — * Pharmaceutical Form: Solution for injection in pre-filled syringe
  * Route of Administration: Subcutaneous use
  * Dose and Administration details :
    2 x 1 mL Certolizumab Pegol at Week 0, followed by
  * 1 x 1 mL Certolizumab Pegol plus 1 x 1 mL Placebo (for blinding reasons) in the Certolizumab Pegol 200 mg arm at Weeks 2, 4, 6, 8 and 10
  * 2 x 1 mL Certolizumab Pegol in the Certolizumab Pegol 400 mg arm at Weeks 2, 4, 6, 8 and 10

SUMMARY:
The primary objective is to assess differences in PASI scores between Week 12 of Study C87040 [NCT00245765] and Week 12 of re-treatment in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject having responded to treatment at Week 12 in study C87040 and having relapsed during the follow-up period
* Female subjects either postmenopausal for at least one year, surgically incapable of childbearing, or effectively practising an acceptable method of contraception.Subjects agreed to continue using adequate contraception during the study and for 12 weeks after the last dose of CDP870

Exclusion Criteria:

* Subjects with erythrodermic, guttate, generalized pustular form of psoriasis
* Any recent serious or life-threatening infection or any current sign or symptom that may indicate an infection (e.g., fever, cough)
* Positive hepatitis B surface antigen test and /or hepatitis C antibody test results
* Positive human immunodeficiency virus (HIV) test result
* White blood cell counts less than 4000 per cubic millimeter or more than 20000 per cubic millimeter
* Suspected or diagnosed demyelinating disease of the central nervous system (e.g. multiple sclerosis or optic neuritis)
* Systemic Lupus Erythematosus
* Participation in a clinical study within the past 3 months except Study C87040
* Any other condition, which in the Investigator's judgment would make the subject unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB Pharma
Locations (14):
- France (5):
  - Besançon
  - Créteil
  - Nice
  - Paris
  - Pierre-Bénite
- Germany (9):
  - Berlin
  - Bonn
  - Essen
  - Frankfurt
  - Hamburg
  - Kiel
  - Mahlow
  - Mainz
  - Münster

REFERENCES:
- [Result] Reich K, Ortonne JP, Gottlieb AB, Terpstra IJ, Coteur G, Tasset C, Mease P. Successful treatment of moderate to severe plaque psoriasis with the PEGylated Fab' certolizumab pegol: results of a phase II randomized, placebo-controlled trial with a re-treatment extension. Br J Dermatol. 2012 Jul;167(1):180-90. doi: 10.1111/j.1365-2133.2012.10941.x. Epub 2012 Jun 11. PMID 22413944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in April 2006 and concluded in May 2007.
Pre-assignment Details: Participant Flow refers to the Intention-to-treat population.
Period: Overall Study
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Started | 34 | 37
Completed | 32 | 35
Not Completed | 2 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Decision of the sponsor | 0 | 1
Not completed — Patient no longer available | 1 | 0
Not completed — Patient relocated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Intention-To-Treat (ITT) population consisting of all enrolled subjects.
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg | Total Title
Number analyzed (Participants) | 34 | 37 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 35 | 69
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.24 (8.64) | 44.57 (12.47) | 44.41 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 23 | 27 | 50

OUTCOME MEASURES:

1. Primary Outcome: Difference in Psoriasis Activity and Severity Index (PASI) Scores Between Week 12 of the First Treatment in Study C87040 [NCT00245765] and Week 12 of Re-treatment in This Study
Description: The PASI is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0=no disease, the maximum score is 72=maximal disease. The difference was calculated by 'PASI score at re-treatment Week 12' minus 'PASI score at First Treatment Week 12'.
Time Frame: Week 12 in C87040 [NCT00245765] and Week 12 in this study
Population: Intention-To-Treat (ITT) population with Last Observation Carried Forward (LOCF).
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
units on a scale | 1.25 [0.10 to 4.40] | 0.20 [0.00 to 0.70]

2. Secondary Outcome: Achievement of a Psoriasis Activity and Severity Index (PASI75) Response at Week 12 of Re-treatment Period From First Treatment Baseline in Study C87040
Description: Determining the PASI score involves the evaluation of erythema, infiltration, and desquamation and body surface area involvement over 4 body regions. These regions are the head, trunk, upper and lower extremities.
  PASI75 response at Week 12 of re-treatment is defined as a decrease in PASI score at Week 12 in this study from Baseline in study C87040 of at least 75 %.
Time Frame: Week 12
Population: Intention-To-Treat (ITT) population.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage of subjects | 67.6 | 86.5

3. Secondary Outcome: Achievement of a Psoriasis Activity and Severity Index (PASI75) Response at Week 12 of Re-treatment Period From Re-treatment Baseline in This Study
Description: Determining the PASI score involves the evaluation of erythema, infiltration, and desquamation and body surface area involvement over 4 body regions. These regions are the head, trunk, upper and lower extremities.
  PASI75 response at Week 12 of re-treatment is defined as a decrease in PASI score at Week 12 in this study from Baseline in this study of at least 75 %.
Time Frame: Week 12
Population: Intention-To-Treat (ITT) population.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage of subjects | 50.0 | 75.7

4. Secondary Outcome: Achievement of a Psoriasis Activity and Severity Index (PASI50) Response at Week 12 of Re-treatment Period From First Treatment Baseline in Study C87040
Description: Determining the PASI score involves the evaluation of erythema, infiltration, and desquamation and body surface area involvement over 4 body regions. These regions are the head, trunk, upper and lower extremities.
  PASI50 response at Week 12 of re-treatment is defined as a decrease in PASI score at Week 12 in this study from Baseline in study C87040 of at least 50 %.
Time Frame: Week 12
Population: Intention-To-Treat (ITT) population.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage of subjects | 76.5 | 89.2

5. Secondary Outcome: Achievement of a Psoriasis Activity and Severity Index (PASI50) Response at Week 12 of Re-treatment Period From Re-treatment Baseline in This Study
Description: Determining the PASI score involves the evaluation of erythema, infiltration, and desquamation and body surface area involvement over 4 body regions. These regions are the head, trunk, upper and lower extremities.
  PASI50 response at Week 12 of re-treatment is defined as a decrease in PASI score at Week 12 in this study from Baseline in this study of at least 50 %.
Time Frame: Week 12
Population: Intention-To-Treat (ITT) population.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage of subjects | 67.6 | 89.2

6. Secondary Outcome: Achievement of a Psoriasis Activity and Severity Index (PASI90) Response at Week 12 of Re-treatment Period From First Treatment Baseline in Study C87040
Description: Determining the PASI score involves the evaluation of erythema, infiltration, and desquamation and body surface area involvement over 4 body regions. These regions are the head, trunk, upper and lower extremities.
  PASI90 response at Week 12 of re-treatment is defined as a decrease in PASI score at Week 12 in this study from Baseline in study C87040 of at least 90 %.
Time Frame: Week 12
Population: Intention-To-Treat (ITT) population.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage of subjects | 35.3 | 48.6

7. Secondary Outcome: Achievement of a Psoriasis Activity and Severity Index (PASI90) Response at Week 12 of Re-treatment Period From Re-treatment Baseline in This Study
Description: Determining the PASI score involves the evaluation of erythema, infiltration, and desquamation and body surface area involvement over 4 body regions. These regions are the head, trunk, upper and lower extremities.
  PASI90 response at Week 12 of re-treatment is defined as a decrease in PASI score at Week 12 in this study from Baseline in this study of at least 90 %.
Time Frame: Week 12
Population: Intention-To-Treat (ITT) population.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage of subjects | 29.4 | 40.5

8. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at First Treatment Baseline in Study C87040
Description: Determining the PASI score involves the evaluation of erythema, infiltration, and desquamation and body surface area involvement over 4 body regions. These regions are the head, trunk, upper and lower extremities.
  The score value ranges from 0 to 72, with higher scores indicating higher Psoriasis activity and severity.
Time Frame: First treatment Baseline in study C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
units on a scale | 20.90 [18.40 to 25.50] | 21.00 [18.30 to 23.60]

9. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 1 of First Treatment Period in Study C87040
Description: as for outcome 8
Time Frame: Week 1 of first treatment Period in study C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 33 | 37
units on a scale | 18.60 [12.60 to 21.80] | 18.60 [15.80 to 20.60]

10. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 2 of First Treatment Period in Study C87040
Description: as for outcome 8
Time Frame: Week 2 of first treatment Period in study C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
units on a scale | 14.00 [10.10 to 18.20] | 14.40 [11.10 to 16.00]

11. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 3 of First Treatment Period in Study C87040
Description: as for outcome 8
Time Frame: Week 3 of first treatment Period in study C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 36
units on a scale | 8.65 [7.20 to 12.60] | 11.35 [8.40 to 13.40]

12. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 4 of First Treatment Period in Study C87040
Description: as for outcome 8
Time Frame: Week 4 of first treatment Period in study C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
units on a scale | 6.55 [5.40 to 10.30] | 8.60 [6.60 to 11.40]

13. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 6 of First Treatment Period in Study C87040
Description: as for outcome 8
Time Frame: Week 6 of first treatment Period in study C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
units on a scale | 4.60 [2.00 to 6.40] | 5.80 [4.40 to 7.50]

14. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 8 of First Treatment Period in Study C87040
Description: as for outcome 8
Time Frame: Week 8 of first treatment Period in study C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
units on a scale | 3.55 [2.20 to 4.70] | 3.80 [2.70 to 5.00]

15. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 10 of First Treatment Period in Study C87040
Description: as for outcome 8
Time Frame: Week 10 of first treatment Period in study C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 36
units on a scale | 2.10 [1.10 to 3.80] | 2.45 [1.40 to 3.60]

16. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 12 of First Treatment Period in Study C87040
Description: as for outcome 8
Time Frame: Week 12 of first treatment Period in study C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
units on a scale | 1.60 [0.90 to 2.70] | 1.80 [1.20 to 2.60]

17. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Re-treatment Baseline in This Study
Description: as for outcome 8
Time Frame: Re-treatment Baseline in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
units on a scale | 14.40 [12.40 to 17.60] | 14.20 [12.90 to 17.50]

18. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 2 of Re-treatment Period in This Study
Description: as for outcome 8
Time Frame: Week 2 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
units on a scale | 10.00 [7.90 to 11.50] | 9.90 [8.20 to 13.20]

19. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 4 of Re-treatment Period in This Study
Description: as for outcome 8
Time Frame: Week 4 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
units on a scale | 6.30 [3.40 to 7.70] | 6.90 [4.30 to 8.90]

20. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 6 of Re-treatment Period in This Study
Description: as for outcome 8
Time Frame: Week 6 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 35
units on a scale | 3.65 [2.50 to 6.40] | 4.40 [2.80 to 5.80]

21. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 8 of Re-treatment Period in This Study
Description: as for outcome 8
Time Frame: Week 8 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 33 | 36
units on a scale | 3.70 [1.40 to 6.00] | 2.70 [1.80 to 4.80]

22. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 10 of Re-treatment Period in This Study
Description: as for outcome 8
Time Frame: Week 10 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 32 | 34
units on a scale | 2.70 [1.20 to 5.80] | 2.25 [1.20 to 3.50]

23. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Week 12 of Re-treatment Period in This Study
Description: as for outcome 8
Time Frame: Week 12 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 32 | 35
units on a scale | 2.80 [1.40 to 6.30] | 2.00 [0.60 to 3.30]

24. Secondary Outcome: Psoriasis Activity and Severity Index (PASI) Score at Last Re-treatment Visit in This Study
Description: as for outcome 8
Time Frame: Last re-treatment visit in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
units on a scale | 3.35 [1.40 to 6.30] | 2.00 [0.60 to 3.30]

25. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 1 of First Treatment Period in C87040
Description: Determining the PASI score involves the evaluation of erythema, infiltration, and desquamation and body surface area involvement over 4 body regions. These regions are the head, trunk, upper and lower extremities.
  The score value ranges from 0 to 72, with higher scores indicating higher Psoriasis activity and severity. A positive value in percentage change from Baseline indicates an improvement from Baseline.
Time Frame: From first treatment Baseline in study C87040 to Week 1 of first treatment Period in C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 33 | 37
percentage change | 12.70 [5.88 to 25.85] | 13.17 [2.34 to 19.09]

26. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 2 of First Treatment Period in C87040
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to Week 2 of first treatment Period in C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage change | 29.94 [13.73 to 46.48] | 31.90 [24.43 to 42.70]

27. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 3 of First Treatment Period in C87040
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to Week 3 of first treatment Period in C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 36
percentage change | 54.99 [40.00 to 66.95] | 50.92 [44.68 to 58.93]

28. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 4 of First Treatment Period in C87040
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to Week 4 of first treatment Period in C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage change | 62.53 [47.47 to 78.83] | 60.31 [50.95 to 67.41]

29. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 6 of First Treatment Period in C87040
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to Week 6 of first treatment Period in C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage change | 80.03 [66.67 to 88.86] | 72.41 [66.67 to 79.55]

30. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 8 of First Treatment Period in C87040
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to Week 8 of first treatment Period in C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage change | 82.80 [73.33 to 93.17] | 84.78 [74.86 to 87.79]

31. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 10 of First Treatment Period in C87040
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to Week 10 of first treatment Period in C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 36
percentage change | 87.74 [82.54 to 96.08] | 89.94 [81.76 to 93.88]

32. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 12 of First Treatment Period in C87040
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to Week 12 of first treatment in C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage of Baseline value
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage of Baseline value | 92.45 [86.73 to 96.51] | 90.60 [89.30 to 95.92]

33. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Re-treatment Baseline in This Study
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to re-treatment Baseline in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage change | 33.48 [26.96 to 38.87] | 32.00 [20.63 to 37.02]

34. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 2 of Re-treatment Period in This Study
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to Week 2 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage change | 58.41 [49.12 to 68.18] | 53.08 [40.14 to 57.33]

35. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 4 of Re-treatment Period in This Study
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to Week 4 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage change | 71.01 [66.37 to 80.98] | 72.56 [62.30 to 79.31]

36. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 6 of Re-treatment Period in This Study
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to Week 6 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 35
percentage change | 80.86 [71.72 to 90.00] | 83.62 [75.91 to 88.41]

37. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 8 of Re-treatment Period in This Study
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to Week 8 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 33 | 36
percentage change | 82.00 [70.59 to 91.53] | 86.46 [76.60 to 91.60]

38. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 10 of Re-treatment Period in This Study
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to Week 10 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 32 | 34
percentage change | 87.13 [77.78 to 96.19] | 90.75 [82.51 to 95.65]

39. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Week 12 of Re-treatment Period in This Study
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to Week 12 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage of Baseline value
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 32 | 35
percentage of Baseline value | 84.11 [76.47 to 95.95] | 91.78 [83.47 to 96.92]

40. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From First Treatment Baseline in Study C87040 to Last Re-treatment Visit in This Study
Description: as for outcome 25
Time Frame: From first treatment Baseline in study C87040 to last re-treatment visit (up to Week 12) in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage change | 83.46 [76.47 to 94.07] | 87.94 [83.47 to 96.30]

41. Secondary Outcome: Percentage Change in Psoriasis Activity and Severity Index (PASI) Score From Re-treatment Baseline in This Study to Week 12 of Re-treatment in This Study
Description: as for outcome 25
Time Frame: From re-treatment Baseline in this study to Week 12 of re-treatment in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage of Baseline value
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 32 | 35
percentage of Baseline value | 78.75 [65.91 to 93.80] | 87.59 [80.00 to 95.88]

42. Secondary Outcome: Best Psoriasis Activity and Severity Index (PASI) Score During the 12 Week First Treatment Period in Study C87040
Description: as for outcome 8
Time Frame: 12 week first treatment Period in study C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
units on a scale | 1.60 [0.80 to 2.70] | 1.60 [0.80 to 2.00]

43. Secondary Outcome: Best Psoriasis Activity and Severity Index (PASI) Score During the 12 Week Re-treatment Period in This Study
Description: as for outcome 8
Time Frame: 12 week re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
units on a scale | 2.00 [1.20 to 4.20] | 1.80 [0.60 to 2.80]

44. Secondary Outcome: Time to Reach Best Psoriasis Activity and Severity Index (PASI) Score During the 12 Week First Treatment Period in Study C87040
Description: as for outcome 8
Time Frame: 12 week first treatment Period in study C87040
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
weeks | 11.00 [10.00 to 12.00] | 12.00 [10.29 to 12.00]

45. Secondary Outcome: Time to Reach Best Psoriasis Activity and Severity Index (PASI) Score During the 12 Week Re-treatment Period in This Study
Description: as for outcome 8
Time Frame: 12 week re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
weeks | 8.00 [6.00 to 10.00] | 9.86 [8.00 to 10.14]

46. Secondary Outcome: Psoriasis Global Assessment (PGA) Rating at Re-treatment Baseline in This Study
Description: The overall severity of the disease was evaluated using the following 6-point scale:
  5 = Severe: Very marked plaque elevation, scaling, and/or erythema. 4 = Moderate to severe: Marked plaque elevation, scaling, and/or erythema. 3 = Moderate: Moderate plaque elevation, scaling, and/or erythema. 2 = Mild: Slight plaque elevation, scaling, and/or erythema
  1 = Almost clear: Intermediate between mild and clear 0 = Clear: No signs of psoriasis (post-inflammatory hyperpigmentation may be present)
Time Frame: Re-treatment Baseline in this study
Population: Intention-To-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
Participants
  Clear | 0 | 0
  Almost clear | 0 | 0
  Mild | 1 | 1
  Moderate | 14 | 13
  Moderate to severe | 15 | 19
  Severe | 4 | 4

47. Secondary Outcome: Psoriasis Global Assessment (PGA) Rating at Week 2 of Re-treatment Period in This Study
Description: as for outcome 46
Time Frame: Week 2 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
Participants
  Clear | 0 | 0
  Almost clear | 0 | 0
  Mild | 9 | 8
  Moderate | 21 | 17
  Moderate to severe | 2 | 9
  Severe | 2 | 3

48. Secondary Outcome: Psoriasis Global Assessment (PGA) Rating at Week 4 of Re-treatment Period in This Study
Description: as for outcome 46
Time Frame: Week 4 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
Participants
  Clear | 1 | 0
  Almost clear | 7 | 8
  Mild | 11 | 11
  Moderate | 13 | 16
  Moderate to severe | 2 | 1
  Severe | 0 | 1

49. Secondary Outcome: Psoriasis Global Assessment (PGA) Rating at Week 6 of Re-treatment Period in This Study
Description: as for outcome 46
Time Frame: Week 6 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
Participants
  Clear | 3 | 4
  Almost clear | 9 | 8
  Mild | 11 | 15
  Moderate | 10 | 5
  Moderate to severe | 1 | 1
  Severe | 0 | 1
  Missing | 0 | 3

50. Secondary Outcome: Psoriasis Global Assessment (PGA) Rating at Week 8 of Re-treatment Period in This Study
Description: as for outcome 46
Time Frame: Week 8 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
Participants
  Clear | 3 | 5
  Almost clear | 9 | 14
  Mild | 10 | 11
  Moderate | 8 | 6
  Moderate to severe | 3 | 0
  Severe | 0 | 0
  Missing | 1 | 1

51. Secondary Outcome: Psoriasis Global Assessment (PGA) Rating at Week 10 of Re-treatment Period in This Study
Description: as for outcome 46
Time Frame: Week 10 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
Participants
  Clear | 7 | 5
  Almost clear | 9 | 15
  Mild | 7 | 11
  Moderate | 6 | 3
  Moderate to severe | 3 | 0
  Severe | 0 | 0
  Missing | 2 | 3

52. Secondary Outcome: Psoriasis Global Assessment (PGA) Rating at Week 12 of Re-treatment Period in This Study
Description: as for outcome 46
Time Frame: Week 12 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
Participants
  Clear | 6 | 10
  Almost clear | 12 | 11
  Mild | 4 | 11
  Moderate | 6 | 1
  Moderate to severe | 3 | 1
  Severe | 1 | 0
  Missing | 2 | 3

53. Secondary Outcome: Psoriasis Global Assessment (PGA) Rating at Last Re-treatment Visit in This Study
Description: as for outcome 46
Time Frame: Last re-treatment visit in this study
Population: Intention-To-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
Participants
  Clear | 6 | 10
  Almost clear | 12 | 13
  Mild | 5 | 12
  Moderate | 7 | 1
  Moderate to severe | 3 | 1
  Severe | 1 | 0

54. Secondary Outcome: Percentage of Subjects Who Achieve a Psoriasis Global Assessment (PGA) Clear or Almost Clear Response at Week 12 of Re-treatment in This Study
Description: as for outcome 46
Time Frame: Week 12 of re-treatment in this study
Population: Intention-To-Treat (ITT) population.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage of subjects | 52.9 | 56.8

55. Secondary Outcome: BSA (Body Surface Area) Affected by Psoriasis at Re-treatment Baseline in This Study
Description: Two methods were used for the evaluation of BSA:
  1. The area of one side of a subject's flat closed hand was used to represent 1 % to the total body surface area (BSA) to estimate the extent of skin involvement in subjects with psoriasis
  2. The rule of nines method assumed that the total BSA comprises head (9 %), anterior trunk (upper, 9 %; lower, 9 %), posterior trunk (upper, 9 %; lower, 9 %), each leg (anterior, 9 %; posterior, 9 %), each arm (9 %) and genitalia (1 %)
Time Frame: Re-treatment Baseline in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage of Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage of Body Surface Area | 16.0 [13.0 to 20.0] | 15.0 [12.0 to 18.0]

56. Secondary Outcome: BSA (Body Surface Area) Affected by Psoriasis at Week 2 of Re-treatment Period in This Study
Description: as for outcome 55
Time Frame: Week 2 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage of Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage of Body Surface Area | 12.5 [10.0 to 17.0] | 14.0 [10.0 to 15.0]

57. Secondary Outcome: BSA (Body Surface Area) Affected by Psoriasis at Week 4 of Re-treatment Period in This Study
Description: as for outcome 55
Time Frame: Week 4 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage of Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage of Body Surface Area | 9.5 [5.0 to 13.0] | 10.0 [6.0 to 14.0]

58. Secondary Outcome: BSA (Body Surface Area) Affected by Psoriasis at Week 6 of Re-treatment Period in This Study
Description: as for outcome 55
Time Frame: Week 6 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage of Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 35
percentage of Body Surface Area | 6.0 [5.0 to 11.0] | 7.0 [5.0 to 11.0]

59. Secondary Outcome: BSA (Body Surface Area) Affected by Psoriasis at Week 8 of Re-treatment Period in This Study
Description: as for outcome 55
Time Frame: Week 8 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage of Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 33 | 36
percentage of Body Surface Area | 5.0 [3.0 to 10.0] | 5.0 [4.0 to 10.0]

60. Secondary Outcome: BSA (Body Surface Area) Affected by Psoriasis at Week 10 of Re-treatment Period in This Study
Description: as for outcome 55
Time Frame: Week 10 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage of Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 32 | 34
percentage of Body Surface Area | 3.0 [2.0 to 7.0] | 4.0 [3.0 to 6.0]

61. Secondary Outcome: BSA (Body Surface Area) Affected by Psoriasis at Week 12 of Re-treatment Period in This Study
Description: as for outcome 55
Time Frame: Week 12 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage of Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 32 | 34
percentage of Body Surface Area | 3.0 [2.0 to 8.0] | 3.0 [1.0 to 5.0]

62. Secondary Outcome: BSA (Body Surface Area) Affected by Psoriasis at Last Re-treatment Visit in This Study
Description: as for outcome 55
Time Frame: Last re-treatment visit in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percentage of Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percentage of Body Surface Area | 3.5 [2.0 to 10.0] | 3.0 [1.0 to 5.0]

63. Secondary Outcome: Change in BSA (Body Surface Area) Score From First Treatment Baseline in C87040 to Re-treatment Baseline in This Study
Description: Two methods were used for the evaluation of BSA:
  1. The area of one side of a subject's flat closed hand was used to represent 1 % to the total body surface area (BSA) to estimate the extent of skin involvement in subjects with psoriasis
  2. The rule of nines method assumed that the total BSA comprises head (9 %), anterior trunk (upper, 9 %; lower, 9 %), posterior trunk (upper, 9 %; lower, 9 %), each leg (anterior, 9 %; posterior, 9 %), each arm (9 %) and genitalia (1 %) A positive value in Change from Baseline indicates an improvement from Baseline. The higher the positive value, the higher the change.
Time Frame: From first treatment Baseline in C87040 to re-treatment Baseline in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percent of total Body Surface Area | 9.0 [3.0 to 11.0] | 7.0 [5.0 to 12.0]

64. Secondary Outcome: Change in BSA (Body Surface Area) Score From First Treatment Baseline in C87040 to Week 2 of Re-treatment Period in This Study
Description: as for outcome 63
Time Frame: From first treatment Baseline in C87040 to Week 2 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percent of total Body Surface Area | 11.0 [9.0 to 15.0] | 10.0 [7.0 to 15.0]

65. Secondary Outcome: Change in BSA (Body Surface Area) Score From First Treatment Baseline in C87040 to Week 4 of Re-treatment Period in This Study
Description: as for outcome 63
Time Frame: From first treatment Baseline in C87040 to Week 4 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percent of total Body Surface Area | 13.0 [10.0 to 17.0] | 12.0 [10.0 to 20.0]

66. Secondary Outcome: Change in BSA (Body Surface Area) Score From First Treatment Baseline in C87040 to Week 6 of Re-treatment Period in This Study
Description: as for outcome 63
Time Frame: From first treatment Baseline in C87040 to Week 6 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 35
percent of total Body Surface Area | 13.5 [12.0 to 20.0] | 19.0 [10.0 to 24.0]

67. Secondary Outcome: Change in BSA (Body Surface Area) Score From First Treatment Baseline in C87040 to Week 8 of Re-treatment Period in This Study
Description: as for outcome 63
Time Frame: From first treatment Baseline in C87040 to Week 8 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 33 | 36
percent of total Body Surface Area | 15.0 [10.0 to 20.0] | 18.0 [14.0 to 26.0]

68. Secondary Outcome: Change in BSA (Body Surface Area) Score From First Treatment Baseline in C87040 to Week 10 of Re-treatment Period in This Study
Description: as for outcome 63
Time Frame: From first treatment Baseline in C87040 to Week 10 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 32 | 34
percent of total Body Surface Area | 15.0 [12.0 to 23.0] | 20.5 [15.0 to 30.0]

69. Secondary Outcome: Change in BSA (Body Surface Area) Score From First Treatment Baseline in C87040 to Week 12 of Re-treatment Period in This Study
Description: as for outcome 63
Time Frame: From first treatment Baseline in C87040 to Week 12 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 32 | 34
percent of total Body Surface Area | 15.0 [12.0 to 23.0] | 20.5 [15.0 to 28.0]

70. Secondary Outcome: Change in BSA (Body Surface Area) Score From First Treatment Baseline in C87040 to Last Re-treatment Visit in This Study
Description: as for outcome 63
Time Frame: From first treatment Baseline in C87040 to last re-treatment visit (up to Week 12) in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percent of total Body Surface Area | 15.0 [12.0 to 19.0] | 22.0 [15.0 to 28.0]

71. Secondary Outcome: Change in BSA (Body Surface Area) Score From Re-treatment Baseline in This Study to Week 2 of Re-treatment Period in This Study
Description: as for outcome 63
Time Frame: From re-treatment Baseline in this study to Week 2 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percent of total Body Surface Area | 2.5 [0.0 to 5.0] | 0.0 [0.0 to 1.0]

72. Secondary Outcome: Change in BSA (Body Surface Area) Score From Re-treatment Baseline in This Study to Week 4 of Re-treatment Period in This Study
Description: as for outcome 63
Time Frame: From re-treatment Baseline in this study to Week 4 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percent of total Body Surface Area | 4.0 [3.0 to 8.0] | 3.0 [2.0 to 4.0]

73. Secondary Outcome: Change in BSA (Body Surface Area) Score From Re-treatment Baseline in This Study to Week 6 of Re-treatment Period in This Study
Description: as for outcome 63
Time Frame: From re-treatment Baseline in this study to Week 6 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 35
percent of total Body Surface Area | 7.0 [4.0 to 11.0] | 7.0 [5.0 to 11.0]

74. Secondary Outcome: Change in BSA (Body Surface Area) Score From Re-treatment Baseline in This Study to Week 8 of Re-treatment Period in This Study
Description: as for outcome 63
Time Frame: From re-treatment Baseline in this study to Week 8 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 33 | 36
percent of total Body Surface Area | 10.0 [3.0 to 12.0] | 9.0 [6.0 to 12.0]

75. Secondary Outcome: Change in BSA (Body Surface Area) Score From Re-treatment Baseline in This Study to Week 10 of Re-treatment Period in This Study
Description: as for outcome 63
Time Frame: From re-treatment Baseline in this study to Week 10 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 32 | 34
percent of total Body Surface Area | 12.5 [5.0 to 14.0] | 9.5 [7.0 to 13.0]

76. Secondary Outcome: Change in BSA (Body Surface Area) Score From Re-treatment Baseline in This Study to Week 12 of Re-treatment Period in This Study
Description: as for outcome 63
Time Frame: From re-treatment Baseline in this study to Week 12 of re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 32 | 34
percent of total Body Surface Area | 10.5 [5.0 to 16.0] | 10.5 [8.0 to 13.0]

77. Secondary Outcome: Change in BSA (Body Surface Area) Score From Re-treatment Baseline in This Study to Last Re-treatment Visit in This Study
Description: as for outcome 63
Time Frame: From re-treatment Baseline in this study to last re-treatment visit in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: percent of total Body Surface Area
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
percent of total Body Surface Area | 10.0 [5.0 to 15.0] | 11.0 [8.0 to 13.0]

78. Secondary Outcome: Time to Withdrawal From the Treatment Due to Lack of Efficacy or Due to AE ('Worsening or Exacerbation of Psoriasis') During the 12 Week Re-treatment Period in This Study
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: During the 12 week re-treatment Period in this study
Population: Intention-To-Treat (ITT) population.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
Number analyzed (Participants) | 34 | 37
days | 56.00 [56.00 to 56.00] | NA [NA to NA] — No values available since none of the subjects in the CZP 400 mg arm withdrew from the treatment due to lack of efficacy or due to AE ('Worsening or Exacerbation of Psoriasis') during the 12 week re-treatment Period in this study.

ADVERSE EVENTS:
Time Frame: Over the 12 week duration of the study.
Description: Averse Events refer to the Safety Population consisting of all subjects who were dispensed medication.
Arm/Group | Certolizumab Pegol (CZP) 200 mg | Certolizumab Pegol (CZP) 400 mg
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/37
Other Adverse Events (participants affected / at risk) | 9/34 | 11/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Certolizumab Pegol (CZP) 200 mg (N=34) | Certolizumab Pegol (CZP) 400 mg (N=37)
Asthenia (General disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 5 | 3
Tonsillitis (Infections and infestations) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days